CLINICAL TRIAL: NCT07019532
Title: A Prospective Cohort Study for Machine Learning-Based Prediction of Anal Fistula Formation After Perianal Abscess Drainage Based on Drainage Setting, Provider Experience, and MRI Interpretation (PRISM)
Brief Title: Machine Learning-Based Risk Stratification for Fistula Formation After Perianal Abscess Drainage
Acronym: PRISM
Status: Not yet recruiting | Type: Observational
Sponsor: Gumushane State Hospital (Other Government)
Responsible Party: Principal Investigator, Kayahan Eyüboğlu, General Surgery Specialist, Gumushane State Hospital
Other Study IDs: FISTUL-ML-01
Record Dates: First submitted 2025-06-05; First posted 2025-06-13 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Perianal Abscess; Anal Fistula
Keywords: Artificial Intelligence; MR Imaging; Colorectal Surgery; Surgical Outcomes; Drainage; Fistula Prediction
MeSH Terms: conditions — Rectal Fistula

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This prospective cohort study investigates the influence of provider experience and drainage location on fistula formation within 6 months following perianal abscess drainage. Additionally, the study explores the role of artificial intelligence (AI)-based interpretation of magnetic resonance (MR) images in early identification of fistula development.

DETAILED DESCRIPTION:
Perianal abscess drainage is a common surgical procedure. However, subsequent fistula formation remains a significant complication. This study aims to determine whether the procedure setting (operating room, emergency department, or outpatient clinic) and the experience level of the performing clinician affect fistula development rates.

Furthermore, the study evaluates the use of AI-assisted analysis of selected MR images to identify early signs of fistula formation. Selected image slices will be labeled based on radiological reports, and a machine learning model will be trained to predict fistula risk. The study will also compare AI-generated interpretations with expert radiologist assessments to validate performance.

The ultimate goal is to create a risk stratification tool to support clinical decision-making in surgical management of perianal abscesses.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18
* First-time perianal abscess
* Surgical drainage performed

Exclusion Criteria:

* Existing anal fistula history
* Crohn's disease
* Immunosuppressive treatment
* Incomplete 6-month follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (≥18 years old) undergoing surgical drainage for their first perianal abscess at a university or state hospital. Participants must not have a history of anal fistula, Crohn's disease, or be under immunosuppressive therapy. Follow-up duration is 6 months after drainage.
Sampling Method: Non-Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Fistula formation within 6 months | 6 months
  Confirmed by clinical exam, surgical findings, or MR imaging

SECONDARY OUTCOMES:
Correlation between drainage location and fistula rate | 6 months
Correlation between provider experience and fistula complexity | 6 months
Diagnostic accuracy of AI-based MR analysis vs radiologist | 6 months

IPD SHARING:
Plan to Share IPD: Yes
De-identified MR images and anonymized patient-level data will be available for collaborative analysis upon request.
Supporting Information: Study Protocol, ICF, CSR